CLINICAL TRIAL: NCT02524600
Title: Technical Performance of a New Cardiac Technology "IQ-SPECT" Applied to SCINTI-CT Myocardial Imaging With 99mTc-Sestamibi in Coronary Patients
Acronym: IQSCINTIMYOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-030
Record Dates: First submitted 2015-08-05; First posted 2015-08-17 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- New Technology "IQ-SPECT" applied to myocardial imaging (Experimental)
  Interventions: Device: myocardial IQ-SPECT imaging applied to scintigraphic imaging; Device: scintigraphic imaging

INTERVENTIONS:
Device: myocardial IQ-SPECT imaging applied to scintigraphic imaging
Device: scintigraphic imaging

SUMMARY:
Cardiological examination is one of the major directions in nuclear medicine for detection of myocardial ischemia in patients with suspected coronary artery disease. In Caen, they constitute 20% of the activity of nuclear medicine. It is evaluating a new versatile innovative technology (IQ-SPECT) for performing rapid nuclear cardiological examinations (4 minutes) and quality on a SCINTI-CT camera for correcting the mitigation. This technical solution IQ-SPECT was made available to the nuclear medicine department in August 2011. To date, apart from the work on heart ghosts and one publication in abstract form in 2009, no other study have been published.

The goal of the study is to study the technical performance of the innovative technology IQ-SPECT during a SCINTI-CT imaging in patients suspected of coronary disease .

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years (except major patients under guardianship)
* free and informed consent signed
* written and spoken French
* beneficiaries of the social security system
* coronary insufficiency detection needed for patients with signs or symptoms suggestive of coronary insufficiency; or in symptomatic patients, but with a high risk of coronary heart disease: diabetes and / or with multiple cardiovascular risk factors and / or having a peripheral vascular disease

Exclusion Criteria:

* Patients with a recent history (<21 days) acute coronary failure (myocardial infarction, unstable angina);
* Patients with an irregular heartbeat, because of the impossibility of achieving a good quality ECG synchronization (atrial fibrillation, ventricular extra-systole or supraventricular over 25% of cardiac cycles);
* Patients with a pacemaker with a permanent electro-drive at rest;
* Patients with non-ischemic heart disease: primitive dilated cardiomyopathy, severe hypertrophic cardiomyopathy, severe valvular cardiomyopathy (aortic stenosis, aortic or mitral leakage grade> 2), congenital heart disease;
* Patients with severe extra-cardiac disease may interfere with treatment decisions (cancer, severe hepatic or renal impairment);
* Major patients under guardianship;
* Pregnant or lactating women;
* Women in age and condition of childbearing;
* Patients unable to understand the purpose of the study.

Cons-indications to physical stress test:

* Uncontrolled heart failure,
* Pulmonary embolism, phlebitis evolution,
* Myocarditis, pericarditis, endocarditis evolving
* Physical disability,
* Thrombus
* Asthma
* contra-indication for exercise testing as dipyridamole:
* Severe Asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Myocardial perfusion binding | baseline
  * 0 = normal fixing ≥70%
  * 1 = slightly reduced mounting 50-69%
  * 2 = moderately less attachment 30-49%
  * 3 = severely diminished attachment 10-20%
  * 4 = no binding <10%

CONTACTS AND LOCATIONS:
Locations (1):
- Service Imagerie Médicale, Caen, CHU, France